CLINICAL TRIAL: NCT06759636
Title: FRIENDS-01：A Multicenter Open-label Randomized Controlled Study on the Treatment of CTIT of the Efficacy and Safety With Romiplostim N01 Compared to Recombinant Human Interleukin-11
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QLMA-CTIT-IIT-101
Record Dates: First submitted 2024-12-29; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: CTIT: Cancer Therapy Induced Thrombocytopenia
MeSH Terms: interventions — Interleukin-11; oprelvekin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Romiplostim N01 (Experimental): 3.0 µg/kg, subcutaneous injection, once a week. Afterwards, refer to the platelet count evaluated during the visit before the next dosing cycle: ① If the platelet count is less than 50×10^9/L, increase by 1-2μg/kg once a week; ② If the platelet count is between 50-99×10^9/L, increase by 1μg/kg once a week. According to platelet count and symptoms, investigators can adjust the dosage to the maximum dosage of 10μg/kg once a week.
  Interventions: Drug: Romiplostim N01
- Recombinant Human Interleukin-11 (Active Comparator): 25-50μg/kg, subcutaneous injection, once a day
  Interventions: Drug: Recombinant Human Interleukin-11 (rhIL-11)

INTERVENTIONS:
Drug: Romiplostim N01 — 3.0 µg/kg, subcutaneous injection, once a week. Afterwards, refer to the platelet count evaluated during the visit before the next dosing cycle: ① If the platelet count is less than 50×10^9/L, increase by 1-2μg/kg once a week; ② If the platelet count is between 50-99×10^9/L, increase by 1μg/kg once a week. According to platelet count and symptoms, investigators can adjust the dosage to the maximum dosage of 10μg/kg once a week.
  Arms: Romiplostim N01
Drug: Recombinant Human Interleukin-11 (rhIL-11) — 25-50μg/kg, subcutaneous injection, once a day
  Arms: Recombinant Human Interleukin-11

SUMMARY:
FRIENDS-01：A Multicenter Open-label Randomized Controlled Study on the Treatment of CTIT of the Efficacy and Safety With Romiplostim N01 Compared to Recombinant Human Interleukin-11

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntarily participate in this study, sign an informed consent form, and strictly complied with the study protocol requirements；
* 2.Age range from 18 to 75 years old，male or female；
* 3.Diagnosed with a malignant tumor by histopathology and/or cytology and is receiving anti-tumor therapy such as chemotherapy, radiotherapy, immunology, and targeting；
* 4.ECOG PS score: 0-2；
* 5.CTIT patients need two platelet tests, two platelet tests should be performed 24 hours apart, and the platelet value should be between 10×10^9/L - 75×10^9/L；
* 6.Estimated survival time during screening is ≥ 12 weeks, and could be treated with current antitumor regimens for at least 1 cycle；
* 7.Subjects of childbearing age agree to take reliable contraceptive measures (including male or female condoms, contraceptive foam, contraceptive gel, contraceptive film, contraceptive cream, contraceptive suppository, abstinence and the placement of intrauterine devices, etc.) throughout the study period; Excluding female participants who have undergone hysterectomy, bilateral salpingectomy, bilateral tubal ligation, or more than 1 year after menopause, as well as male participants who have undergone bilateral salpingectomy or ligation；
* 8.Adequate organ and bone marrow function.

Exclusion Criteria:

* 1. Platelet values at screening or baseline were ≤10×10^9/L；
* 2.Participants with a history of any hematological malignancy，including but not limited to leukemia, primary immune thrombocytopenia, myeloproliferative diseases, multiple myeloma, and myelodysplastic syndrome；
* 3.Participants had a history of chronic platelet or bleeding disorders，or screening for thrombocytopenia caused by causes other than CIT within the first 6 months, including but not limited to chronic liver disease, splenic hyperfunction, infection, and bleeding；
* 4.Bone marrow invasion or metastasis;
* 5.Have received pelvic and spinal radiation therapy, as well as bone field radiation therapy, or are currently/expected to receive radiation therapy within the three months prior to screening;
* 6.Brain tumors or brain metastases;
* 7.Screening for a history of severe cardiovascular disease within the first 6 months, such as congestive heart failure (NYHA heart function score III-IV), known arrhythmias that increase the risk of thromboembolism, such as atrial fibrillation, after coronary stent implantation, angioplasty, and coronary artery bypass grafting;
* 8.Any history of arterial or venous thrombosis occurring within the first 6 months of screening;
* 9.Screening for clinical manifestations of severe bleeding within the first two weeks, such as gastrointestinal or central nervous system bleeding;
* 10.Neutrophil absolute value < 1.0 × 10^9/L, hemoglobin < 80g/L, allowing the use of granulocyte colony-stimulating factors and red blood cells that comply with clinical norms EPO infusion therapy
* 11.Significant abnormalities in liver function: patients without liver metastasis, ALT/AST>3ULN (upper limit of normal value), TBIL>3ULN； Patients with liver metastasis are present, ALT/AST≥5ULN，TBIL≥5ULN;
* 12.Renal dysfunction: blood creatinine ≥ 1.5ULN or eGFR ≤ 60 ml/min (Cockcroft Gault formula);
* 13.Within the first month prior to screening, patients who have received treatment with thrombopoietin receptor agonists or recombinant human thrombopoietin (rhTPO) or recombinant human interleukin-11 (rhIL-11);
* 14.Received platelet transfusion within the first two weeks of randomization;
* 15.Participants who are known or expected to be allergic or intolerant to Roxetine N01 or rhIL-11 excipients;
* 16.HIV infected individuals;
* 17.Pregnant or lactating women;
* 18.Participants had medically known hereditary prethrombotic syndromes (e.g., clotting factor V Leiden mutation, prothrombin G20210A mutation, or hereditary antithrombin III (ATIII) deficiency);
* 19.Participants were given a vitamin K antagonist within 7 days prior to screening (permitted drugs included low molecular weight heparin, Factor Xa inhibitors, or thrombin inhibitors);
* 20.As assessed by the investigators, the participants had any concomitant medical history that could compromise the participants' safe completion of the study, such as unstable angina, renal failure on hemodialysis, or an active infection requiring intravenous antibiotics;
* 21.Participated in any clinical study of any other investigational drug or device three months prior to screening;
* 22.The researchers believe that participating in the trial poses a significant risk to the health or safety of the subjects, or other circumstances that may affect the efficacy evaluation;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-01-21 (Estimated); Primary Completion 2026-04-21 (Estimated); Study Completion 2026-07-21 (Estimated)

PRIMARY OUTCOMES:
The median number of days when the platelet count reaches 100×10^9/L or the absolute platelet count increases by 50×10^9/L | through study completion, an average of 5 months

SECONDARY OUTCOMES:
The median number of days for patients with baseline PLT counts less than 50×10^9/L and less than 75×10^9/L to achieve a PLT count of 100×10^9/L | through study completion, an average of 5 months
The median number of days in which thrombocytopenia increases from Grade 3 or 4 to Grade 1 or 2 | through study completion, an average of 5 months
The average number of days when the platelet count reaches 100×10^9/L or the absolute platelet count increases by 50×10^9/L | through study completion, an average of 5 months
Proportion of patients with PLT reaching 100×10^9/L or absolute platelet count increase of 50×10^9/L after 1 week of treatment | Within 1 weeks after receiving treatment
Proportion of patients with PLT reaching 100×10^9/L or absolute platelet count increase of 50×10^9/L after 2 weeks of treatment | Within 2 weeks after receiving treatment
Proportion of patients with PLT reaching 100×10^9/L or absolute platelet count increase of 50×10^9/L after 3 weeks of treatment | Within 3 weeks after receiving treatment
Proportion of patients with PLT reaching 100×10^9/L or absolute platelet count increase of 50×10^9/L after 4 weeks of treatment | Within 4 weeks after receiving treatment
Thrombocytopenia level in X+1 cycle of antitumor therapy | through study completion, an average of 5 months
Proportion of bleeding patients | through study completion, an average of 5 months
The incidence of platelet transfusion | through study completion, an average of 5 months
The absolute increase in platelet count after the medication was discontinued | through study completion, an average of 5 months
Effect of Romiplostim N01 on hemoglobin and leukocyte | through study completion, an average of 5 months
Adverse events (evaluated using the Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0), laboratory tests, vital signs, electrocardiograms, and physical examinations, etc | through study completion, an average of 5 months
The incidence and severity of bleeding events ( being evaluated using the WHO Bleeding Scale) should be closely monitored for participants' drug allergies, cardiovascular adverse events, risk of thrombosis, and rhIL-11 related adverse events | through study completion, an average of 5 months

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No